CLINICAL TRIAL: NCT06311409
Title: Validation Study of the Speedy Meyer Fall Scale for Determining the Fall Risk of the Paediatric Patient
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Daniele Ciofi, Princiapl Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: SMFS2019
Record Dates: First submitted 2024-02-23; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Fall Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fall prevention is an essential element in ensuring safe care for paediatric patients. The first step in building a risk reduction programme is the adoption of an assessment tool to identify those most at risk at an early stage. From October 2014 to date, a study has been conducted for the linguistic-cultural validation of the Humpty Dumpty Fall Scale (HDFS) in the Italian context, through a multicentre survey with the help of the Clinical Risk Management Group of the Region of Tuscany.

The objective of this study is the validation of the new Humpty Dumpty Fall Scale defined as Speedy Meyer-Fall Scale (SMFS) by assessing the comprehension and validity of the scale and items via Content Validity Index (SCVI and ICVI) estimation of inter-item reliability (Crombach's alpha), inter-rater reliability (Cohen's K), sensitivity, specificity, PPV, NPV and ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* children admitted as in-patients for whom the parents have given consent to the study, aged between 12 months and 16 years, of any gender, pathology and reason for admission.

Exclusion Criteria:

* not signed consent form

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children admitted as in-patients for whom the parents have given consent to the study, aged between 12 months and 16 years, of any gender, pathology and reason for admission. Population i
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
validation of the SMFS t | through study completion, an average of 1 year
  validation of the SMFS through the assessment of the comprehensibility of the SMFS, the validity of the SMFS through Content Validity Index at item (ICVI) and scale (SCVI) level, and the reliability of the SMFS through inter-item reliability (Cronbach's alpha) and Inter-rater Reliability (Cohen's K)

SECONDARY OUTCOMES:
identification of patients high risk of falls | through study completion, an average of 1 year
  estimation of the sensitivity, specificity, Positive Predictive Value (PPV), Negative Predictive Value (NPV) and ROC curve in clinical practice and their comparison with the theoretical data of the scale in question in order to identify patients at high risk of falls in a paediatric hospital

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Ciofi, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (3):
- Italy (3):
  - AUSL Toscana Sud Est, Arezzo
  - Meyer Children's Hospital IRCCS, Florence
  - Fondazione Gabriele monasterio - Ospedale Pediatrico Apuano Massa, Massa